CLINICAL TRIAL: NCT05124795
Title: Dose Escalation Study to Evaluate the Safety, Tolerability, and Anti-Tumor Activity of Single Agent IMU-935 in Patients With Progressive, Metastatic Castration Resistant Prostate Cancer
Brief Title: IMU-935 in Patients With Progressive, Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Immunic AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P1-IMU-935-CRPC
Record Dates: First submitted 2021-10-29; First posted 2021-11-18 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Castration Resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IMU-935 - low dose, administered twice daily (Experimental): main treatment phase of 3 cycles of 28 days; followed by extended treatment cycles for patients that show clinical benefit from treatment
  Interventions: Drug: IMU-935
- IMU-935 - medium dose, administered twice daily (Experimental): main treatment phase of 3 cycles of 28 days; followed by extended treatment cycles for patients that show clinical benefit from treatment
  Interventions: Drug: IMU-935
- IMU-935 - high dose, administered twice daily (Experimental): main treatment phase of 3 cycles of 28 days; followed by extended treatment cycles for patients that show clinical benefit from treatment
  Interventions: Drug: IMU-935

INTERVENTIONS:
Drug: IMU-935 — IMU-935 capsules

SUMMARY:
Dose escalation study to evaluate the safety, tolerability and anti-tumor activity of single agent IMU-935 in patients with progressive, metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is an open-label, non-randomized Phase 1 dose escalation, followed by dose expansion, study to define the safety, tolerability, biomarker change and anti-tumor activity of IMU-935 in patients with mCRPC. Throughout the study, safety, anti-tumor activity, biomarkers and IMU-935 plasma concentrations will be evaluated at regular intervals as per schedule of assessments. Disease progression will be assessed as per standard medical practice.

The dose escalation and expansion parts of the study will have the same treatment duration with similarly structured treatment cycles.

The study will consist of the following periods:

* Screening Period: Approximately 28 days
* Treatment Phase:

Main treatment over 3 cycles of 28 days each, extended treatment as long as patient benefits

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Male patients with histologically or cytologically confirmed adenocarcinoma of the prostate with no evidence of small cell or neuroendocrine features
* Metastatic disease with limited therapeutic options, prior treatment with at least one next-generation hormonal agent (e.g., abiraterone, enzalutamide, apalutamide, darolutamide) and one taxane line of treatment is allowed
* Progressive disease is defined as rising prostate-specific antigen (PSA) levels ≥2ng/mL and/or radiographic progression according to Prostate Cancer Working Group 3 (PCWG3) criteria at screening
* Able and willing to comply with all study requirements for the duration of the study
* Patients must sign an ICF prior to the start of any study-related procedures

Exclusion Criteria:

* Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy) within 28 days prior to starting study treatment
* Uncontrolled intercurrent illness such as active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with the study protocol
* Malignancy within the previous 2 years with a ≥30% probability of recurrence within 12 months, with the exception of non-melanoma skin cancer or superficial bladder cancer
* Patients receiving strong inhibitors or inducers of cytochrome P450 (CYP) 3A4
* Chronic use of systemic steroid therapy (>1 month of >10 mg prednisone per day or equivalent, except replacement therapy)
* Patients for whom biopsies cannot be taken or are not willing to undergo biopsies
* Positive hepatitis B virus (HBV) surface antigen, hepatitis B core antibody, positive hepatitis C virus (HCV) antibody, and/or HIV-antigen-antibody test at screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence and the grade (severity) of dose-limiting toxicities (DLTs) within 28 days after start of study treatment to identify the MTD and the RP2D | Within 28 days after start of study treatment
  DLTs are abnormal laboratory parameters or adverse events (per National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events V5.0) occurring during the DLT observation period of 28 days from treatment start, assessed as toxicities being related to IMU-935.
Number and severity of adverse events (AEs) reported according to the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | 6 months
  Incidence and severity of adverse events as assessed by CTCAE Version 5.0.

SECONDARY OUTCOMES:
Proportion of patients considered responders to IMU-935 related to decline in prostate specific antigen (PSA) level | 6 months
  Patients with a serum prostate specific antigen (PSA) level decline of ≥30% from their pre-treatment level will be considered responders.
Proportion of patients considered responders to IMU-935 related to decline in circulating tumor cells (CTC) numbers | 6 months
  Patients showing a conversion of circulating tumor cells (CTC) from ≥5 cells/7.5 mL blood at Cycle 1 Day 1 (pre-dose) to ≤4 cells/7.5 mL blood will be considered responders.
Proportion of patients considered responders to IMU-935 related to the objective response based on the Response Evaluation Criteria in Solid Tumors (RECIST) V 1.1 | 6 months
  Response rate as per RECIST V 1.1 will be evaluated centrally to identify responders.

CONTACTS AND LOCATIONS:
Overall Officials: J. B., MD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- Institute of Cancer Research, London, United Kingdom